CLINICAL TRIAL: NCT00231634
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study of the Efficacy and Safety of Topiramate in the Treatment of Obese, Type 2 Diabetic Patients Inadequately Controlled on Sulfonylurea Therapy
Brief Title: A Study of the Efficacy and Safety of Topiramate in Obese, Type 2 Diabetic Patients Inadequately Controlled on Sulfonylurea Therapy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Program discontinued
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR002251
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-01

CONDITIONS: Obesity; Diabetes Mellitus, Type 2; Diabetes Mellitus, Adult-Onset
Keywords: Obesity; Type 2 Diabetes Mellitus; HbA1c; Sulfonylurea; Topiramate; Adult-Onset Diabetes Mellitus (AODM)
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2 | interventions — Topiramate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: topiramate

SUMMARY:
The purpose of this study is to compare the effectiveness and safety of topiramate with placebo in the treatment of obesity and Type 2 diabetes mellitus in patients who have failed on sulfonylurea therapy.

DETAILED DESCRIPTION:
Topiramate is a medication for the treatment of seizures, but not approved for the treatment of obesity. This is a randomized, double-blind, placebo controlled study to evaluate the effectiveness and safety of topiramate in Type 2 diabetic patients with obesity who have failed on treatment with sulfonylurea. After a 4-week enrollment phase and 8-week titration phase, patients receive either topiramate (96, 192, or 256 mg twice daily) or placebo for 44 weeks, followed by a 6-week follow-up phase. Assessments of effectiveness include body weight, hemoglobin type A1c [HbA1c] (a measurement of average blood sugar level over several months), Body Mass Index (BMI), fasting plasma glucose (FPG) level, fasting lipid profile, fasting insulin, uric acid level, blood pressures, and health related quality of life (HRQOL) measures. Safety evaluations, including incidence and severity of adverse events, hypoglycemic episodes, clinical laboratory results such as the liver enzymes, and vital signs, are performed throughout the study. The study hypothesis is that topiramate will be effective in the treatment of type 2 diabetes through weight reduction. During the initial 8-weeks, oral doses taken twice daily of topiramate or placebo will be gradually increased to target doses (either 96 milligrams[mg], 192mg, or 256mg daily); the dose will be maintained for 44 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Type 2 Diabetes, receiving only second generation sulfonylurea therapy (may include: glipizide, gliclazide, glimepiride, glibenclamide/glyburide, and gliquadone) for at least 4 months and on stable dose for at least 2 months
* Body Mass Index >= 27 and < 50
* HbA1c < 11% at enrollment
* Diagnosed hypertension or hyperlipidemia must be controlled
* Female patients must be postmenopausal for at least 1 year, surgically incapable of childbearing, practicing an acceptable method of contraception (requires negative pregnancy test)

Exclusion Criteria:

* Known contraindication or hypersensitivity to topiramate or sulfonylurea therapy
* Pregnancy or women who are nursing or plan to become pregnant during the study
* Diagnosed with Type 1 diabetes
* History of severe or recurrent hypoglycemic episodes
* Treatment with any antidiabetic agent other than sulfonylurea

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2001-05; Study Completion 2002-11 (Actual)

PRIMARY OUTCOMES:
Percent change in body weight and change in Hemoglobin A1c (HbA1c) from baseline to Week 52.

SECONDARY OUTCOMES:
Change from baseline to Week 52 in BMI, FPG; safety evaluations (adverse events, hypoglycemic events) throughout study.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A Study of the Efficacy and Safety of Topiramate in Obese Type 2 Diabetic Patients Inadequately Controlled on Sulfonylurea Therapy — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=465&filename=CR002251_CSR.pdf